CLINICAL TRIAL: NCT00200694
Title: Anti-Proteinuric Response to ACEI, ARB and Diuretics Combination.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: difficulty in patients's inclusion
Sponsor: Nantes University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: BRD 03-5-D
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2009-02-04 (Estimated); Status verified 2009-02

CONDITIONS: Heavy Proteinuria
Keywords: Proteinuria; ACEI; ARB; diuretics; blood pressure; renal failure
MeSH Terms: conditions — Proteinuria; Renal Insufficiency | interventions — Ramipril; Valsartan

INTERVENTIONS:
Drug: ramipril 5 mg + valsartan 80 mg/day,
Drug: ramipril 10 mg + valsartan 160 mg/day,
Drug: ramipril 5 mg + valsartan 80 mg/day + increased dosage of furosémide.

SUMMARY:
Determine the best strategy for proteinuria lowering in patients with proteinuria > 1 g/day receiving ACEI and ARB combination: either increase of ACEI and ARB dosage or increase of diuretic dosage.

ELIGIBILITY:
Inclusion Criteria:

* proteinuria > 1 g/day with ramipril 5 + valsartan 80 mg/day for 2 months
* proteinuria changes < 50% on 3 separate dosages over 2 months.

Exclusion criteria:

* age < 18 or > 80 years systolic BP < 110 or ≥ 140 mmHg, serum creatinine > 250 mmole/L
* serum creatinine increase on ramipril + valsartan > 20%
* intolerance to ACEI or ARB

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18
Dates: Start 2005-03; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent LM Esnault, MD PHD, Principal Investigator — Nantes University Hospital
Locations (1):
- CHU de Nantes, Nantes, France